CLINICAL TRIAL: NCT06282484
Title: A Study on the Relationship Between Gastric Xanthoma and Gastric Cancer and Precancerous Lesions
Status: Completed | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator, Clinical Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: KY20232348-C-1
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gastric Xanthoma; Helicobacter Pylori Infection; Gastric Cancer; Intestinal Metaplasia; Precancerous Lesions
Keywords: gastric cancer; helicobacter pylori; precancerous lesion; Gastric Xanthoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- chronic gastritis: patients with chronic non-atrophic gastritis and chronic atrophic gastritis according to histopathological results
- precancerous lesion: patients with gastric intestinal metaplasia and intraepithelial neoplasia according to histopathological results
- gastric cancer: patients with gastric cancer according to histopathological results

SUMMARY:
To explore the effects of gastric xanthoma on gastric cancer and its precancerous lesions, so as to better prevent the occurrence and development of gastric cancer.

DETAILED DESCRIPTION:
This is a large-scale single center case-control study. Patients were consecutively enrolled and divided into gastric cancer group, gastric precancerous lesions group, and chronic gastritis group, according to histopathological results.Record the location and quantity of gastric xanthoma and situation of Helicobacter pylori infection in each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 75 years old, regardless of gender;
2. Endoscopic/pathological diagnosis: chronic non atrophic gastritis/chronic atrophic gastritis/intestinal metaplasia/dysplasia Hyperplasia/gastric cancer
3. Voluntarily sign an informed consent form.

Exclusion Criteria:

1. Previously underwent upper gastrointestinal surgery
2. Previous diagnosis of malignant tumors
3. Individuals who are unable to cooperate with the questionnaire survey due to mental disorders or other reasons
4. Those who cannot be observed by endoscopy due to acute upper gastrointestinal bleeding or other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing upper gastrointestinal endoscopy at Xijing Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1260 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
corelation between the gastric xanthoma and gastric mucosa diseases | up to 6 months
  we evaluate the corelation between the gastric xanthoma and gastric mucosa diseases according to the histopathological results and the scales the patients finished

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, PhD, Study Director — Xijing Hosipital of Digestive Disease
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No